CLINICAL TRIAL: NCT03232762
Title: Effects of Diet on Pregnancy Outcome and Child Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-00694
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy Related; Diet Modification; Obesity; Hypertension; Pre-Eclampsia; Blood Pressure; Breast Feeding; Birth Weight
MeSH Terms: conditions — Obesity; Hypertension; Pre-Eclampsia; Breast Feeding; Birth Weight | interventions — Whole Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet A (Active Comparator): high proportion of calories from refined grains as a carbohydrate source
  Interventions: Dietary Supplement: Refined Grains
- Diet B (Active Comparator): a high proportion of calories from whole grains
  Interventions: Dietary Supplement: Whole Grains

INTERVENTIONS:
Dietary Supplement: Refined Grains — In week one each patient will have a text message or phone call to report on her diet and the information will be recorded as an attempt to assure compliance.
  Arms: Diet A
Dietary Supplement: Whole Grains — In week one each patient will have a text message or phone call to report on her diet and the information will be recorded as an attempt to assure compliance.
  Arms: Diet B

SUMMARY:
The purpose of the study is to compare 3 different diets in pregnancy, equal in calories, and fats, different in refined grains compared to whole grains as a source of carbohydrates, and in calories from carbohydrate, compared to protein as a source of calories.The hypothesis is that there will be differences in the specified outcomes because the proportions of macronutrients are significant. The primary objective is to detect differences in weight gain.

DETAILED DESCRIPTION:
There will be randomized sequential assignment of pregnant women at the initial clinic visit to Diet A, a high proportion of calories from refined grains as a carbohydrate source, and Diet B, a high proportion of calories from whole grains. Random number assignment is impractical for counseling purposes and blinding not possible. Therefore, randomization by diet assignment by day of initial visit via random number was chosen. If the random number is odd Diet A would be selected, if the random number is even Diet B will be selected for that day.

ELIGIBILITY:
Inclusion Criteria:

* All normal pregnant patients who will be more than three months from term

Exclusion Criteria:

* Illness making it a high risk pregnancy
* Chronic renal disease
* Malignancy
* Congestive heart failure
* Diabetes
* Hypertension

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All will be pregnant women
Enrollment: 303 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

PRIMARY OUTCOMES:
Differences in weight gain | 6 Months

SECONDARY OUTCOMES:
Pre-Term Birth Rate | 6 Months
Neonatal Weight | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Young, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Sun H, Yamada P, Paetow A, Chan M, Arslan A, Landberg R, Dominguez-Bello MG, Young BK. A randomized controlled trial of the effects of whole grains versus refined grains diets on the microbiome in pregnancy. Sci Rep. 2022 May 7;12(1):7509. doi: 10.1038/s41598-022-11571-4. PMID 35525865